CLINICAL TRIAL: NCT02705807
Title: An Open Label, Single-arm Study Evaluating a New Thermostable Formulation of FLOLAN™ in Japanese Subjects With Pulmonary Arterial Hypertension (PAH)
Brief Title: Evaluation of a New Thermostable Formulation of FLOLAN in Japanese Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201614
Record Dates: First submitted 2016-02-25; First posted 2016-03-11 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-01

CONDITIONS: Cardiovascular Disease
Keywords: Pulmonary Arterial Hypertension (PAH); safety; FLOLAN; New Thermostable Formulation; dose adjustment; reformulated diluents; currently marketed diluent
MeSH Terms: conditions — Cardiovascular Diseases; Pulmonary Arterial Hypertension | interventions — Epoprostenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLOLAN arm (Experimental): Subjects will receive the existing FLOLAN treatment (i.e., FLOLAN injection prepared with the currently marketed diluent) for a run-in period of a maximum of 4 weeks, the thermostable formulation of FLOLAN injection (i.e., FLOLAN injection prepared with the reformulated diluent) for a 4-week treatment period and there will be a one-week follow-up visit.
  Interventions: Drug: FLOLAN injection with currently marketed diluent; Drug: FLOLAN injection with reformulated diluent

INTERVENTIONS:
Drug: FLOLAN injection with currently marketed diluent — FLOLAN injection (epoprostenol 0.5 or 1.5) prepared with the currently marketed diluent (epoprostenol sodium+ powder of hydrogen [pH] 10.2 - 10.8 diluent) for Injection.
Drug: FLOLAN injection with reformulated diluent — FLOLAN injection (epoprostenol 0.5 or 1.5) prepared with the reformulated diluent (epoprostenol sodium + pH 11.7 - 12.3 diluent) for Injection.

SUMMARY:
This study is a Phase IV, open-label, single-arm study to assess the safety and the necessity of dose adjustment after switching to FLOLAN injection prepared with the reformulated diluent in Japanese patients with PAH who are receiving higher doses of FLOLAN injection than in other countries. The objective is to evaluate the safety and tolerability of the thermostable formulation of FLOLAN injection (that is [i.e.], FLOLAN injection prepared with the reformulated diluent) when switched from the existing FLOLAN injection treatment (i.e., FLOLAN injection prepared with the currently marketed diluent). The study will include a screening visit, a run-in period of a maximum of 4 weeks with the existing FLOLAN treatment (i.e., FLOLAN injection prepared with the currently marketed diluent), a 4-week treatment period with the thermostable formulation of FLOLAN injection (i.e., FLOLAN injection prepared with the reformulated diluent) and a one-week follow-up visit. Adequate number of subjects will be enrolled in the study in order to have 10 subjects to complete assessments at 4 weeks, including at least 5 subjects as a subset of subjects who consent to undergo right heart catheterisation (RHC) over 24-hour and at Week 4. FLOLAN is a registered trademark of the GlaxoSmithKline [GSK] group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 to 75 years at the time of screening;
* Subjects must be on FLOLAN therapy for pulmonary arterial hypertension (PAH) as approved in the product label;
* Subjects must receive FLOLAN therapy at 45 nanograms (ng)/kilogram (kg)/minute (min) or higher;
* Subjects must be on stable doses of their existing FLOLAN treatment for a minimum of one month prior to screening; it is acceptable to adjust within 10% of dose during the last one month period;
* Subjects must be on stable doses of any current PAH treatments other than FLOLAN therapy in the last 30 days prior to screening;
* Subjects who meet any of the following: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative [serum or urine] human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

  * Non-reproductive potential defined as: Pre-menopausal females with any of the following: documented tubal ligation, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy, or documented bilateral oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
  * Reproductive potential and agrees to follow one of the options listed below in the GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of thermostable formulation of FLOLAN therapy until completion of the follow-up visit.
* Subject must agree not to participate in a clinical study involving another investigational drug or device throughout this study;
* Subjects must be competent to understand the information given in the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved informed consent form and must sign the form prior to the initiation of any study procedures.

Exclusion Criteria:

* Subjects who are given FLOLAN therapy for a condition or in a manner that is outside the approved indication.
* Subjects with congestive heart failure arising from severe left ventricular dysfunction.
* Subjects, with or without supplemental oxygen, who have a resting arterial oxygen saturation (SaO2) <90% as measured by pulse oximetry at screening.
* Subjects have been hospitalised as an emergency or visited the emergency room for a condition related to PAH or treatment for PAH in the last 3 months.
* The subject's clinical condition is such that they are not expected to remain clinically stable for the duration of the study.
* Female subjects who are pregnant or breastfeeding.
* Subjects who have demonstrated noncompliance with previous medical regimens.
* Subjects who have a history of abusing alcohol or illicit drugs within 1 year.
* Subjects who have participated in a clinical study involving another investigational drug or device within four weeks before screening.
* Any concurrent condition that would affect the safety of the subject or in the opinion of the investigator (or subinvestigator) it is not in the best interest of the patient to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Okayama, Japan

REFERENCES:
- [Derived] Mihara K, Ogawa A, Matsubara H, Terao T, Ichikawa Y. Investigation of safety and efficacy of the new more thermostable formulation of Flolan (epoprostenol) in Japanese patients with pulmonary arterial hypertension (PAH)-An open-label, single-arm study. PLoS One. 2018 Apr 2;13(4):e0195195. doi: 10.1371/journal.pone.0195195. eCollection 2018. PMID 29608587

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted a screening visit, a Run-in period of a maximum of 30 days observation, a 4-week treatment period with the thermostable formulation of FLOLAN, and a one-week follow-up visit.
Pre-assignment Details: Ten participants (par.) who gave consent and passed the screening assessments were enrolled in the Run-in period. After the Run-in period, par. underwent Baseline assessments and were switched to thermostable formulation of FLOLAN. All par. underwent right heart catheterisation (RHC) up to 24 hours and at Week 4 after switching to study treatment.
Groups:
- FLOLAN With New Diluent: Japanese par. with pulmonary arterial hypertension (PAH) received FLOLAN prepared with the current marketed diluent (epoprostenol sodium + Potential of Hydrogen [pH] 10.2-10.8 diluent) for Injection in run-in period for a maximum of 30 days, and then switched to FLOLAN prepared with new diluent (epoprostenol sodium + pH 11.7-12.3 diluent) for Injection for 4-weeks in the treatment period. Par. received dose of 47.6 to 113.8 nanogram per kilogram per minute (ng/kg/min) during the treatment period.
Period: Overall Study
Arm/Group | FLOLAN With New Diluent
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.8 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, important medical events which may require medical or surgical interventions. Intention-to-Treat (ITT) population: comprised of all participants who have received at least one dose of the thermostable formulation of FLOLAN.
Time Frame: Up to Week 4
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Participants
  Any AE | 2
  Any Drug-Related AE | 1
  Any SAE | 0

2. Primary Outcome: Number of Participants With Mild, Moderate or Severe AEs
Description: Intensity for an AE and SAE is categorized as mild if an event is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities; moderate if an event is sufficiently discomforting to interfere with normal everyday activities; severe if that prevents normal everyday activities.
Time Frame: Up to Week 4
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Participants
  Mild, Nausea | 1
  Mild, Hepatic function abnormal | 1

3. Primary Outcome: Percentage of Basophils, Eosinophils, Lymphocytes, Monocytes, and Total Neutrophils in Blood at Baseline and Week 4
Description: Blood samples were collected for the measurement of percentage of basophils, eosinophils, lymphocytes, monocytes, and total neutrophils in blood at Baseline (BL) and Week 4 (W4). The Baseline values are those collected within 0.5 hour (hr) prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Percentage
  Basophils BL | 0.61 (0.331)
  Basophils W4 | 0.45 (0.321)
  Eosinophils BL | 2.66 (1.789)
  Eosinophils W4 | 3.25 (3.221)
  Lymphocytes BL | 22.87 (4.181)
  Lymphocytes W4 | 22.37 (6.453)
  Monocytes BL | 5.16 (1.766)
  Monocytes W4 | 4.46 (1.710)
  Total Neutrophils BL | 68.70 (6.134)
  Total Neutrophils W4 | 69.47 (8.623)

4. Primary Outcome: Absolute Values of Hemoglobin at Baseline and Week 4
Description: Blood samples were collected for measurement of hemoglobin values at Baseline (BL) and Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: Gram/Liter (G/L)
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Gram/Liter (G/L)
  BL | 135.5 (13.37)
  W4 | 124.1 (10.31)

5. Primary Outcome: Absolute Values of Hematocrit at Baseline and Week 4
Description: Blood samples were collected for measurement of hematocrit values at Baseline (BL) and Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Liter (L)
  BL | 0.3969 (0.03230)
  W4 | 0.3662 (0.02682)

6. Primary Outcome: Absolute Values of Platelet Count and White Blood Cell Count at Baseline and Week 4
Description: Blood samples were collected for measurement of platelets and white blood cells (WBC) at Baseline (BL) and Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: Giga/Liter (GI/L)
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Giga/Liter (GI/L)
  Platelet count, BL | 181.9 (75.46)
  Platelet count, W4 | 153.4 (51.58)
  WBC count, BL | 0.0065 (0.00125)
  WBC count, W4 | 0.0063 (0.00140)

7. Primary Outcome: Absolute Values of Red Blood Cell Count at Baseline and Week 4
Description: Blood samples were collected for measurement of red blood cells at Baseline (BL) and Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: terabinary/liter (Ti/L))
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
terabinary/liter (Ti/L))
  BL | 0.0482 (0.00357)
  W4 | 0.0446 (0.00344)

8. Primary Outcome: Absolute Values of Albumin and Total Protein at Baseline and Week 4
Description: Blood samples were collected for measurement of albumin and total protein at Baseline (BL) and Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
G/L
  Albumin, BL | 43.8 (6.03)
  Albumin, W4 | 41.1 (2.64)
  Total protein, BL | 68.0 (7.27)
  Total protein, W4 | 63.9 (4.51)

9. Primary Outcome: Absolute Values of Total and Direct Bilirubin, Creatinine, and Uric Acid at Baseline and Week 4
Description: Blood samples were collected for measurement of total and direct bilirubin, creatinine (CRT), and uric acid (UA) at Baseline (BL) and Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Micromoles per liter
  Total Bilirubin, BL | 9.063 (2.9120)
  Total Bilirubin, W4 | 8.550 (3.2244)
  Direct Bilirubin, BL | 0.855 (0.9012)
  Direct Bilirubin, W4 | 1.368 (1.0815)
  CRT, BL | 58.1672 (7.19132)
  CRT, W4 | 50.4764 (8.28689)
  UA, BL | 349.1476 (93.83901)
  UA, W4 | 313.4596 (70.10066)

10. Primary Outcome: Absolute Values of Alanine Aminotransferase, Aspartate Aminotransferase, Alkaline Phosphatase, Gamma Glutamyltransferase, Lactate Dehydrogenase and Creatine Kinase at Baseline and Week 4
Description: Blood samples were collected for measurement of Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP), Gamma Glutamyltransferase (GGT), Lactate Dehydrogenase (LDH) and Creatine Kinase (CK) at Baseline (BL) and Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
International units per liter (IU/L)
  ALT, BL | 15.9 (7.56)
  ALT, W4 | 19.6 (21.71)
  AST, BL | 14.0 (3.89)
  AST, W4 | 16.4 (11.35)
  ALP, BL | 181.0 (57.02)
  ALP, W4 | 175.2 (69.45)
  GGT, BL | 22.7 (17.46)
  GGT, W4 | 22.1 (17.69)
  LDH, BL | 165.2 (33.77)
  LDH, W4 | 160.8 (34.81)
  CK, BL | 40.8 (15.13)
  CK, W4 | 44.7 (17.22)

11. Primary Outcome: Absolute Values of Urea/Blood Urea Nitrogen, Glucose, Chloride, Sodium, Potassium, Magnesium, Phosphorus (Inorganic), and Calcium at Baseline and Week 4
Description: Blood samples were collected for measurement of urea/Blood Urea Nitrogen (Urea/BUN), glucose, chloride, sodium, potassium, magnesium, phosphorus, inorganic, and calcium at Baseline (BL) and Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: Millimoles per litre (mmol/L)
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Millimoles per litre (mmol/L)
  Urea/BUN, BL | 4.6767 (1.07034)
  Urea/BUN, W4 | 4.4625 (0.99917)
  Glucose, BL | 4.9959 (0.34814)
  Glucose, W4 | 5.7675 (2.05053)
  Chloride, BL | 103.8 (4.64)
  Chloride, W4 | 103.9 (4.01)
  Sodium, BL | 139.6 (1.96)
  Sodium, W4 | 138.0 (1.76)
  Potassium, BL | 3.61 (0.373)
  Potassium, W4 | 3.56 (0.255)
  Magnesium, BL | 0.8467 (0.06767)
  Magnesium, W4 | 0.7891 (0.03242)
  Phosphorus, inorganic, BL | 1.2399 (0.15686)
  Phosphorus, inorganic, W4 | 1.1947 (0.19553)
  Calcium, BL | 2.2380 (0.13100)
  Calcium, W4 | 2.1357 (0.07174)

12. Primary Outcome: Absolute Values of Free Triiodothyronine and Free Thyroxine at Baseline and Week 4
Description: Blood samples were collected for measurement of Free Triiodothyronine (FT3) and Free Thyroxine (FT4) at Baseline (BL) and Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: picomoles per litre (pmol/L)
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
picomoles per litre (pmol/L)
  FT3, BL | 5.0974 (1.26044)
  FT3, W4 | 4.9280 (0.47048)
  FT4, BL | 14.6847 (3.46426)
  FT4, W4 | 14.2857 (2.47336)

13. Primary Outcome: Absolute Values of Thyroid Stimulating Hormone at Baseline and Week 4
Description: Blood samples were collected for measurement of Thyroid Stimulating Hormone (TSH) at Baseline (BL) and Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: milliunits per litre (mU/L)
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
milliunits per litre (mU/L)
  TSH, BL | 2.426 (4.4045)
  TSH, W4 | 1.822 (2.5287)

14. Primary Outcome: Number of Participants With the Indicated Urinalysis Findings
Description: Urine protein, urine glucose, and occult blood were assessed at Baseline (BL) and Week 4 (W4). Dipstick test was performed for routine urinalysis. Abnormal values such as trace, 1+, 2+, 3+ and positive have been reported. The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline').
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Participants
  Urine glucose, BL, Trace | 0
  Urine glucose, BL, 1+ | 0
  Urine glucose, BL, 2+ | 0
  Urine glucose, BL, 3+ | 0
  Urine glucose, BL, Positive | 0
  Urine glucose, W4, Trace | 0
  Urine glucose, W4, 1+ | 0
  Urine glucose, W4, 2+ | 0
  Urine glucose, W4, 3+ | 0
  Urine glucose, W4, Positive | 0
  Urine occult blood, BL, Trace | 2
  Urine occult blood, BL, 1+ | 1
  Urine occult blood, BL, 2+ | 0
  Urine occult blood, BL, 3+ | 0
  Urine occult blood, BL, Positive | 0
  Urine occult blood, W4, Trace | 0
  Urine occult blood, W4, 1+ | 1
  Urine occult blood, W4, 2+ | 0
  Urine occult blood, W4, 3+ | 0
  Urine occult blood, W4, Positive | 0
  Urine protein, BL, Trace | 5
  Urine protein, BL, 1+ | 1
  Urine protein, BL, 2+ | 0
  Urine protein, BL, 3+ | 0
  Urine protein, BL, Positive | 0
  Urine protein, W4, Trace | 2
  Urine protein, W4, 1+ | 0
  Urine protein, W4, 2+ | 0
  Urine protein, W4, 3+ | 0
  Urine protein, W4, Positive | 0

15. Primary Outcome: Number of Participants With the Indicated Electrocardiogram (ECG) Findings
Description: A safety 12-lead ECG was performed at Baseline (BL), 24 hr after switching to the new Flolan diluent and Week 4 (W4). Any abnormal clinically significant (CS) and not clinically significant (NCS) findings were reported. ECG abnormaility with respect to CS and NCS findings were judged by the investigator. The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Baseline, 24 hour and Week 4
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Participants
  BL, NCS | 9
  BL, CS | 1
  24 hr, NCS | 9
  24 hr, CS | 1
  W4, NCS | 10
  W4, CS | 0

16. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured at Baseline, 1 hr, 3 hr, 24 hr, Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline'). Change from Baseline is defined as the difference between the post-dose visit value and the Baseline value.
Time Frame: Baseline, 1 hour, 3 hour, 24 hour and Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Millimeters of mercury (mmHg)
  SBP, 1 hr | 4.2 (5.77)
  SBP, 3 hr | 1.2 (7.73)
  SBP, 24 hr | 1.1 (10.17)
  SBP, Week 4 | 2.1 (8.12)
  DBP, 1 hr | -0.6 (8.06)
  DBP, 3 hr | 0.7 (5.52)
  DBP, 24 hr | 0.9 (6.98)
  DBP, Week 4 | 2.5 (8.03)

17. Primary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured at Baseline, 1 hr, 3 hr, 24 hr, Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline'). Change from Baseline is defined as the difference between the post-dose visit value and the Baseline value.
Time Frame: Baseline and up to Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Beats per minute (bpm)
  1 hr | 1.4 (11.57)
  3 hr | 2.3 (11.54)
  24 hr | 5.1 (9.27)
  Week 4 | 4.0 (9.76)

18. Primary Outcome: Change From Baseline in Body Weight
Description: Body weight was measured at Baseline (BL) and Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline'). Change from Baseline is defined as the difference between the post-dose visit value and the Baseline value. Participants with body weight outside and within the clinical concern reference range (<50kg) has been presented.
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Participants
  > clinical concern range, BL | 0
  < clinical concern range, BL | 6
  > clinical concern range, W4 | 0
  < clinical concern range, W4 | 6

19. Primary Outcome: Absolute Values of Oxygen Saturation
Description: Oxygen saturation was measured by pulse oximetry at Baseline (BL), 1 hr, 3 hr, 24 hr, Week 4 (W4). The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline').
Time Frame: Baseline and up to Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Percentage
  BL | 97.6 (0.70)
  1 hr | 98.0 (1.15)
  3 hr | 97.6 (1.51)
  24 hr | 97.7 (1.16)
  Week 4 | 97.8 (1.55)

20. Secondary Outcome: Number of Events to Adjust Dose of FLOLAN Based on the Change From Baseline to 3 Hours in Mean Pulmonary Artery Pressure (mPAP)
Description: To assess the frequency of dose adjustment requirements based on the changes from baseline in mPAP up to 3 hours after dosing.The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline'). Participants who gave consent to undergo right heart catheterisation (RHC) over 24-hour and at week 4 were assessed. Change from Baseline is defined as the difference between the post-dose visit value and the Baseline value.
Time Frame: Up to Week 4
Population: ITT population
Measure: Number; unit: Number of events
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Number of events
  Yes | 0
  No | 10

21. Secondary Outcome: Number of Participants With the Reason for the Change Dose of the Thermostable Formulation of FLOLAN
Description: All reasons for FLOLAN dose adjustments after the switch were listed.
Time Frame: Up to Week 4
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Participants
  Adverse event | 0
  Other | 2

22. Secondary Outcome: Change From Baseline in N-terminal Pro B-type Natriuretic Peptide (NT Pro BNP)
Description: Blood samples were collected at Baseline, 24 hours after the first dose of thermostable formulation of FLOLAN, and Week 4 for measurement of NT pro BNP. The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline'). Change from Baseline is defined as the difference between the post-dose visit value and the Baseline value.
Time Frame: Baseline and up to Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: nanogram/liter
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
nanogram/liter
  24 hr | -1.8 (21.14)
  Week 4 | 33.7 (103.66)

23. Secondary Outcome: Number of Participants in Each World Health Organization (WHO) Functional Class
Description: The WHO functional classes of PAH range from Class I (without limitation in physical activity) to Class IV (inability to perform a physical activity without any symptoms).
Time Frame: Baseline and Week 4
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Participants
  WHO Class I, BL | 1
  WHO Class II, BL | 9
  WHO Class III, BL | 0
  WHO Class IV, BL | 0
  WHO Class I, W4 | 0
  WHO Class II, W4 | 10
  WHO Class III, W4 | 0
  WHO Class IV, W4 | 0

24. Secondary Outcome: Number of Participants With Change of WHO Functional Class From Previous Visit
Description: WHO Functional Classification of physical activity limitations: I (no limitation) and IV (unable to carry out any physical activity without symptoms). The change from baseline in WHO class was classified as Improved (decrease in functional class), No Change (functional class stayed the same), and Deteriorated (functional class increased). The change from baseline in WHO functional class at Week 4 has been presented in the table. The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline')
Time Frame: Up to Week 4
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
Participants
  Improved | 0
  Deteriorated | 1
  No change | 9

25. Secondary Outcome: Change From Baseline in Mean Pulmonary Arterial Pressure (mPAP) and Mean Right Atrial Pressure (mRAP)
Description: mPAP and mRAP are hemodynamic parameters. The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline'). Change from Baseline is defined as the difference between the post-dose visit value and the Baseline value.
Time Frame: Baseline and up to Week 4
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
mmHg
  mPAP, 1hr | 0.5 (2.17)
  mPAP, 3hr | 1.5 (3.66)
  mPAP, 24hr | -0.5 (3.41)
  mPAP, Week4 | 1.9 (2.96)
  mRAP, 1hr | -0.9 (2.42)
  mRAP, 3hr | -0.1 (3.07)
  mRAP, 24hr | 0.3 (3.89)
  mRAP, Week4 | 1.5 (3.06)

26. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resist (PVR)
Description: The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline'). Change from Baseline is defined as the difference between the post-dose visit value and the Baseline value.
Time Frame: Baseline and up to Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: millimeter mercury/liter/minute
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
millimeter mercury/liter/minute
  1hr | 0.204 (2.2976)
  3hr | -0.077 (0.9716)
  24hr | 0.196 (1.2514)
  Week 4 | 0.368 (1.5393)

27. Secondary Outcome: Change From Baseline in Cardiac Output (CO)
Description: Cardiac output is the volume of blood pumped by the heart per minute. The Baseline values are those collected within 0.5 hr prior to the first dose of the new diluent formulation ('Visit 2 - Baseline'). Change from Baseline is defined as the difference between the post-dose visit value and the Baseline value.
Time Frame: Baseline and up to Week 4
Population: ITT population
Measure: Mean (Standard Deviation); unit: liter/minute
Arm/Group | FLOLAN With New Diluent
Number analyzed (Participants) | 10
liter/minute
  1hr | -0.070 (1.2320)
  3hr | 0.460 (1.1843)
  24hr | -0.020 (0.8854)
  Week 4 | 0.408 (0.9700)

ADVERSE EVENTS:
Time Frame: AEs and SAEs will be collected from the start of treatment with the thermostable formulation of FLOLAN until the follow-up contact (approximately up to Day 65).
Description: SAEs and non-serious AEs were collected in Intention-to-Treat (ITT) population, comprising of all participants who have received at least one dose of the thermostable formulation of FLOLAN.
Arm/Group | FLOLAN With New Diluent
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLOLAN With New Diluent (N=10)
Nausea (Gastrointestinal disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.